CLINICAL TRIAL: NCT00295984
Title: Treatment of Classical Kaposi Sarcoma With Nicotine Dermal Patch: A Phase II Trial
Brief Title: Nicotine Skin Patch in Treating Patients With Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000462444; NCI-06-C-N033; NCT00339755 (obsolete NCT alias)
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2006-08

CONDITIONS: Sarcoma
Keywords: classic Kaposi sarcoma; recurrent Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Kaposi | interventions — Nicotine

INTERVENTIONS:
Drug: nicotine

SUMMARY:
RATIONALE: Nicotine may stimulate the immune system to kill Kaposi's sarcoma cells.

PURPOSE: This phase II trial is studying the side effects and how well the nicotine skin patch works in treating patients with Kaposi's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the toxicity and efficacy of transdermal nicotine applied to lesions in patients with classic Kaposi's Sarcoma.

OUTLINE: This is a double-blind, placebo-controlled study.

Patients apply a nicotine dermal patch to a selected lesion and a placebo patch to the other lesion, replacing the same type of fresh patch every other day, during the first 2 weeks, increasing the nicotine dose in week 3 and again in week 5 for a total of 15 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven classic Kaposi's sarcoma (KS)
* At least 2 KS lesions that can be measured (minimum diameter 0.5 cm to maximum diameter 3 cm) and located on body sites (leg, arm, torso, dorsum of foot or hand) to which a patch can be applied

  * A third measurable lesion (if available) of the same size can be located on any body site
* KS lesions must be separated by at least 8.0 cm at their centers and 6.0 cm at closest edges
* Patient must be a nonsmoker

  * No smoking, chewing, or other use of tobacco within the past year

PATIENT CHARACTERISTICS:

* HIV antibody negative
* Willing to shower or bathe no more than every other day
* No life-threatening conditions
* Not pregnant
* Fertile patients must use effective contraception
* Chronic conditions (e.g., hypertension or diabetes) must be stable and well controlled
* No history of HIV/AIDS, unstable angina pectoris, or claudication
* ECOG performance status 0-1

PRIOR CONCURRENT THERAPY:

* No prior biopsy of the selected KS lesion(s) within the past 90 days
* No prior systemic therapy for KS within the past 90 days
* No concurrent systemic or local conventional treatment for KS
* No prior use of a nicotine product within the past year
* No prior surgery, chemotherapy, biologic therapy, or radiotherapy within the past 90 days
* No prior organ allograft

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-03; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Tumor response at weeks 9 and 15

CONTACTS AND LOCATIONS:
Overall Officials: James J. Goedert, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Goedert JJ, Scoppio BM, Pfeiffer R, Neve L, Federici AB, Long LR, Dolan BM, Brambati M, Bellinvia M, Lauria C, Preiss L, Boneschi V, Whitby D, Brambilla L. Treatment of classic Kaposi sarcoma with a nicotine dermal patch: a phase II clinical trial. J Eur Acad Dermatol Venereol. 2008 Sep;22(9):1101-9. doi: 10.1111/j.1468-3083.2008.02720.x. Epub 2008 Apr 1. PMID 18384551